CLINICAL TRIAL: NCT02046668
Title: A Randomised Placebo Controlled Trial. The Effect of Spironolactone on Pain in Older People With Osteoarthritis
Brief Title: The Effect of Spironolactone on Pain in Older People With Osteoarthritis
Acronym: SPIR-OA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13/WS/0232; 2013-002638-19 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis of knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- spironolactone (Active Comparator): 25mg spironolactone daily
  Interventions: Drug: spironolactone
- Placebo (Placebo Comparator): Matched Placebo
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — spironolactone 25mg daily for 12 weeks
  Other Names: Aldactone

SUMMARY:
This pilot study will obtain preliminary evidence on which to base sample size calculations for a future trial of whether spironolactone (an aldosterone blocker) reduces knee pain in older people with symptomatic OA knee when given in addition to usual analgesia. Aldosterone is known to be pro-inflammatory, and spironolactone suppresses cytokine production in chronic arthritis. This application builds on previous work by the applicants showing that spironolactone significantly improved quality of life (particularly pain) in frail older people. The investigators will recruit 86 people (aged 70 years or over) with well-defined OA knee to 25mg spironolactone daily or to matching placebo for 12 weeks. The primary outcome is the between group difference in change in WOMAC pain sub-score at 12 weeks. Secondary outcomes are the WOMAC stiffness and physical function subscales and health related quality of life (EQ-5D). Morning cortisol levels will be measured to assess the effect of mineralocorticoid receptor blockade on glucocorticoid levels, which may mediate the anti-inflammatory effect of spironolactone; and urinary CTX-II, and serum matrix metalloproteinase-3 (MMP-3) will be measured as biomarkers as both are sensitive to the effects of pharmacological interventions for osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent
2. Community dwelling
3. Aged 70 years and over
4. Symptomatic idiopathic OA knee according to American College of Rheumatology clinical and radiographic criteria (ie Knee pain - with or without crepitus and presence of osteophytes on x ray)
5. To avoid floor effects, participants will require to have moderate (or more severe) pain at screening in at least 2 out of 5 WOMAC pain score items
6. To have been in receipt (prescription or/and over the counter) of one or more analgesic agents at a therapeutic dose for at least 2 months
7. Willing to have knee x-ray if one has not been taken in preceding 12 months

Exclusion Criteria:

1. Clinical diagnosis of symptomatic heart failure
2. History of inflammatory arthritis
3. Already taking spironolactone
4. Previous intolerance to spironolactone
5. Known allergies to spironolactone or lactose
6. Objection to taking capsules made from animal sourced gelatine
7. Taking oral NSAIDs (because of the increased risk of renal impairment when combined with spironolactone)
8. Taking ACE inhibitors or ARBs (angiotensin II receptor antagonists). ARBs have many properties similar to those of ACE inhibitors. Both will be exclusion because of the increased risk of acute kidney injury and hyperkalaemia, and because our previous study also excluded those on ACE inhibitors (and ARBs) and treatment was safe and well tolerated.
9. Supine hypotension (supine systolic blood pressure <100mmHg at screening)
10. Significant chronic kidney disease (eGFR<40ml/min)
11. Serum sodium<130mmol/l
12. Serum potassium>5.0mmol/l
13. Symptomatic orthostatic hypotension (measured at screening)
14. Nursing home resident
15. Wheelchair bound
16. Participating in another clinical trial (other than observational trials and registries) concurrently or within 30 days prior to screening for entry into this study
17. Known contraindication to spironolactone therapy
18. Participant who is terminally ill, defined as less than 3 months expected survival

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Between group difference in change in WOMAC pain subscale (5 items) | 12 weeks

SECONDARY OUTCOMES:
Between group difference in change in WOMAC stiffness subscale. | 12 weeks

OTHER OUTCOMES:
Between group difference in change in WOMAC physical function subscales. | 12 weeks
Between group difference in change in health-related quality of life measured by EQ-5D questionnaire. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marion ET McMurdo, MBChB, MD, Study Director — University of Dundee; Miles Witham, BM BCh, MRCP, Principal Investigator — University of Dundee; Vera Cvoro, Mb CHB, MRCP, Principal Investigator — NHS Fife
Locations (2):
- United Kingdom (2):
  - NHS Fife, Kirkcaldy, Fife
  - NHS Tayside, Dundee, Tayside

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/26413749